CLINICAL TRIAL: NCT04930016
Title: Quality of Life and Survival of Patients With Colorectal Cancer 5 Years After Surgery and Their Aftercare Situation During the COVID-19 Pandemic - Long-term Follow-up of the Randomized Trial DIQOL
Brief Title: Quality of Life and Survival of Patients With Colorectal Cancer 5 Years After Surgery - Follow-up of the RCT DIQOL
Acronym: DIQOLFollow-up
Status: Completed | Type: Observational
Sponsor: Tumor Center Regensburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Monika Klinkhammer-Schalke, Director of the Tumor Center Regensburg, Tumor Center Regensburg
Other Study IDs: DIQOL_Follow-up_2021
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Quality of Life; Colorectal Cancer; Colorectal Neoplasms; Survivorship
Keywords: quality of life; colorectal cancer; complex intervention; survivorship; health services research
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Former DIQOL intervention group: In the present follow-up study no interventions are administered. This group encompasses patients who had been part of the intervention group of the completed RCT DIQOL with the following intervention: Patients answered QoL questionnaires after surgery and at 3, 6, 12, and 18 months postoperatively. Results were transferred to a QoL-profile consisting of 13 QoL scales. Three experts with various professional background used the individual patient's QoL-profile and clinical and sociodemographic information to generate a QoL-report including therapy recommendations which was sent to the patient's doctor. Specific therapeutic options for the treatment of QoL had been defined: pain therapy, psychotherapy, social support, nutrition counseling, stoma care, physiotherapy, and fitness.
  Interventions: Behavioral: Quality of life diagnosis and therapy during the completed RCT DIQOL
- Former DIQOL control group: In the present follow-up study no interventions are administered. This group encompasses patients who had been part of the control group of the completed RCT DIQOL: Patients answered QoL questionnaires after surgery and at 3, 6, 12, and 18 months postoperatively but their doctor neither received a QoL-profile nor a QoL-report.

INTERVENTIONS:
Behavioral: Quality of life diagnosis and therapy during the completed RCT DIQOL — Quality of life measurement, diagnosis, and tailored therapy (pain therapy, psychotherapy, social support, nutrition, stoma care, physiotherapy, fitness)
  Groups: Former DIQOL intervention group

SUMMARY:
This observational follow-up study of the randomized trial (RCT) DIQOL investigates long-term effects of an intervention with quality of life (QoL) diagnosis and therapy on present QoL, survival, and recurrence-free survival of colorectal cancer survivors more than 5 years after surgery.

Moreover, patients' experiences with aftercare for colorectal cancer during the COVID-19 pandemic and their recollections of their illness and therapy are examined.

DETAILED DESCRIPTION:
In a complex intervention a clinical pathway with quality of life (QoL) diagnosis and tailored therapy had been developed for patients with colorectal cancer and its effectiveness was evaluated in a randomized trial (RCT DIQOL, NCT02321813, Klinkhammer-Schalke et al, 2020). In the RCT DIQOL a total of 220 patients were randomised (1:1) into two groups: a care pathway, including QoL-profiles consisting of 13 QoL scales plus specific therapeutic recommendations forwarded to the patient's doctor (intervention) or standard postoperative care (control). QoL was measured (EORTC QLQ-C30, QLQ-CR29) in all patients after surgery and during aftercare (3, 6, 12, 18 months postoperatively). A need for QoL therapy was defined as a score <50 points on at least one QoL scale. It was demonstrated that the proportion of patients with a need for QoL therapy was significantly lower in intervention group patients at 12 months after surgery (primary endpoint).

Until now, it is unclear whether there are also long-term benefits of QoL diagnosis and therapy. Therefore, the aim of this observational, cross-sectional follow-up study of the RCT DIQOL is to investigate long-term effects of the intervention on present QoL (EORTC QLQ-C30, QLQ-CR29), overall survival, and recurrence-free survival more than 5 years after surgery by comparing former intervention and control group patients. Moreover, participants will be asked for their experiences during aftercare in relation of the COVID-19 pandemic and for their recollection of their illness and therapy. Data are collected via questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* former participants of the RCT DIQOL with a primary diagnosis of colorectal cancer between 01/2014 and 10/2015 who did not refuse to participate during the RCT
* informed consent

Exclusion Criteria:

- none -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Former participants of the RCT DIQOL with a primary diagnosis of colorectal cancer between 01/2014 and 10/2015 who had been surgically treated in one of four participating certified centers for colorectal cancer (Krankenhaus Barmherzige Brüder Regensburg, Germany; Caritas-Krankenhaus St. Josef Regensburg, Germany; Klinikum Neumarkt, Germany; Klinikum St. Elisabeth Straubing, Germany). Originally, 220 patients were included in the RCT DIQOL. Of the 220 participants who were included in the RCT 12 patients refused participation during the trial so that the final sample for the follow-up study encompasses 208 patients. The questionnaire is mailed to survivors of this cohort. Overall survival and recurrence-free surival will be analzyed in all 208 former study participants.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
need for QoL therapy of colorectal cancer survivors | >5 years after surgery for colorectal cancer
  proportion of patients in both groups with a need for QoL therapy (<50 points in at least one dimension) more than 5 years after surgery
specific need for QoL therapy of colorectal cancers survivors in specific QoL dimensions | >5 years after surgery for colorectal cancer
  rates of patients with a need for QoL therapy in each single dimension of the QoL-profile more than 5 years after surgery

SECONDARY OUTCOMES:
overall survival | surgery for colorectal cancer (01/2014-10/2015) up to 10/2021
  survival after surgery for colorectal cancer
recurrence-free survival | surgery for colorectal cancer (01/2014-10/2015) up to 10/2021
  recurrence-free survival after surgery for colorectal cancer
aftercare of colorectal cancer survivors during the COVID-19 pandemic | >5 years after surgery for colorectal cancer
  self-created questionnaire with quantitative questions asking whether and how the COVID-19 pandemic affected ´aftercare
colorectal cancer survivors' recollections of their illness an therapy | >5 years after surgery for colorectal cancer
  self-created questionnaire with three qualitative questions asking for worst experiences during the colorectal cancer episode, positive aspects of the illness, and any advice survivors would give to newly diagnosed patients

CONTACTS AND LOCATIONS:
Overall Officials: Monika Klinkhammer-Schalke, MD, Prof., Study Chair — Tumor Center Regensburg; Patricia Lindberg-Scharf, PhD, Principal Investigator — Tumor Center Regensburg
Locations (1):
- Tumor Center Regensburg, Institute of Quality Management and Health Services Research of the University of Regensburg, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD that underlie the results in a publication are planned to be made available upon request of scientists.
Time Frame: 6 months after date of publication until 60 months after date of publication
Access Criteria: Data will be made available to other scientists upon request for nonprofit research. The contact address is monika.klinkhammer-schalke@ur.de. Scientists are required to send their predefined statistical analysis plan. Together with the scientific review board of the Tumor Center Regensburg a decision will be made based on the quality and usefulness of planned statistical analysis. In case of a positive decision the scientist is required to sign a contract for data usage before receiving anonymized IPD.

REFERENCES:
- [Background] Klinkhammer-Schalke M, Steinger B, Koller M, Zeman F, Furst A, Gumpp J, Obermaier R, Piso P, Lindberg-Scharf P; Regensburg QoL Study Group. Diagnosing deficits in quality of life and providing tailored therapeutic options: Results of a randomised trial in 220 patients with colorectal cancer. Eur J Cancer. 2020 May;130:102-113. doi: 10.1016/j.ejca.2020.01.025. Epub 2020 Mar 13. PMID 32179445
- [Derived] Volkel V, Steinger B, Koller M, Klinkhammer-Schalke M, Lindberg-Scharf P. Colorectal cancer survivors' long-term recollections of their illness and therapy up to seven years after enrolment into a randomised controlled clinical trial. BMC Cancer. 2023 Feb 13;23(1):149. doi: 10.1186/s12885-023-10604-z. PMID 36782134